CLINICAL TRIAL: NCT05783869
Title: Effect of Cardiovascular Comorbidities on Disease Severity and Quality of Life in Patients With Acute Exacerbation of Non-cystic Fibrosis Bronchiectasis
Brief Title: Study of Bronchiectasis and Associated Cardiovascular Comorbidities
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: Aliae AR Mohamed Hussein [ahussein (Unknown)
Responsible Party: Principal Investigator, Ahmad Shaddad, Lecturer of pulmonary medicine Assuit university, Assiut University
Other Study IDs: 23455668
Record Dates: First submitted 2023-02-12; First posted 2023-03-24 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Echocardiography; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with bronchiectasis and cardiovascular comorbidities: Patients with Bronchiectasis had no comorbidities other than cardiovascular comorbidities during the study period.
  Interventions: Device: Echocardiography
- Patients with bronchiectasis and without cardiovascular comorbidities: Patients with Bronchiectasis had no comorbidities.
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography — echocardiographic study of both groups
  Other Names: Pulmonary function test; Routine laboratory investigations and inflammatory markers

SUMMARY:
Effect of cardiovascular comorbidities on disease severity and quality of life in Patients with acute exacerbation of non-cystic fibrosis bronchiectasis

DETAILED DESCRIPTION:
The study will include patients with bronchiectasis, and in an attempt to correlate the effect and burden of cardiovascular comorbidities in those patients, we will study the quality of life in those patients in comparison to the control group ( patients with bronchiectasis and without any other comorbidities) using SF-36 quality of life questionnaire. We will also study the inflammatory markers in both groups using D-dimer, BNP, and CRP and correlate them with the frequency of hospital admission, the severity of symptoms, and the general health state.

ELIGIBILITY:
Inclusion Criteria:

• Any Patients with Bronchiectasis had no comorbidities other than cardiovascular comorbidities during the study period.

Exclusion Criteria:

* Any Patients who refuse to participate in the study.
* Any other comorbidity or end-organ failure may affect the study's result.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients at the study period attending the chest department at Assuit university
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
assessment of BNP (Brain natriuretic peptide) pg/ml levels in patients with bronchiectasis and cardiovascular comorbidities. | March 2023 to September 2023
  Serum BNP (Brain natriuretic peptide) pg/ml will be compared in both groups.
Assessment of Quality of life in patients and control groups using The Short Form (36) Health Survey (SF-36) | March 2023 to September 2023
  The Short Form (36) Health Survey will be performed in both groups. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

SECONDARY OUTCOMES:
Hospitalization frequency in patient group compared to control group. | March 2023 to September 2023
  Number of hospital admission in the last year will be compared in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Shaddad, Principal Investigator — Assuit University Faculty of Medicine; Ahmad Shaddad, Principal Investigator — Assiut University Faculty of Medicine
Locations (1):
- Assiut unviresty - Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided